CLINICAL TRIAL: NCT02686086
Title: Chronic Obstructive Pulmonary Disease (COPD) Lung Volume and Symptom Scores Following Bronchodilator Therapy Administration by Vibrating Mesh and Standard Jet Nebulisers: A Pilot Comparison Study
Brief Title: A Pilot Comparison Study of Vibrating Mesh Versus Standard Jet Nebuliser for Bronchodilator Delivery in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor of Medicine, Beaumont Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beaumont
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard hospital jet nebuliser (Placebo Comparator): Patients admitted to hospital with an acute exacerbation of COPD and prescribed nebulised bronchodilator therapy (combined short-acting salbutamol 2.5mg and ipratropium 0.5mg) will receive their prescribed medication via a standard hospital jet nebuliser.
  Spirometry, lung volume measurement and symptom score (Borg breathlessness scale) will be recorded pre-nebulisation and at one hour post-nebulisation.
  Interventions: Device: Standard hospital jet nebuliser; Drug: Combined salbutamol 2.5 mg and ipratropium 0.5mg nebule
- Vibrating mesh nebuliser (Active Comparator): Patients admitted to hospital with an acute exacerbation of COPD and prescribed nebulised bronchodilator therapy (combined short-acting salbutamol 2.5mg and ipratropium 0.5mg) will receive their prescribed medication via a vibrating mesh nebuliser (Aerogen Solo) rather than the standard hospital nebuliser Spirometry, lung volume measurement and symptom score (Borg breathlessness scale) will be recorded pre-nebulisation and at one hour post-nebulisation.
  Interventions: Device: vibrating mesh nebuliser; Drug: Combined salbutamol 2.5 mg and ipratropium 0.5mg nebule

INTERVENTIONS:
Device: vibrating mesh nebuliser — The Aerogen Solo vibrating mesh nebuliser is an approved 13 485 class II medical device (CE marked) nebuliser licenced for the delivery of physician-prescribed medications for inhalation which are approved for use with a general purpose nebuliser. It has been shown in previous laboratory and clinical studies to have superior drug delivery to standard jet nebulisers.
  Arms: Vibrating mesh nebuliser
Device: Standard hospital jet nebuliser — The "standard hospital jet nebuliser" refers to the nebuliser in clinical use currently throughout Beaumont Hospital and used for the administration of nebulised medications
  Arms: Standard hospital jet nebuliser
Drug: Combined salbutamol 2.5 mg and ipratropium 0.5mg nebule — All patients admitted to hospital with an exacerbation of COPD are administered nebulised bronchodilators (salbutamol 2.5mg/ipratropium 0.5mg combination) as standard of care

SUMMARY:
Treatment of chronic obstructive pulmonary disease (COPD) incorporates various modes of inhalation therapy. The response to treatments is dose dependent thus applying the most efficient device to administer the treatment is integral. Evaluation of the efficacy of nebulisation devices in the treatment of COPD is limited. Technological development in recent years has led to new devices that optimize lung deposition and reduce the time needed for treatment.

The aim of this study is to compare the vibrating mesh and jet nebuliser methods of delivering bronchodilator medication to patients hospitalised with an acute exacerbation of COPD, with respect to lung function and efficacy in spontaneously breathing patients.

DETAILED DESCRIPTION:
Treatment of chronic obstructive pulmonary disease (COPD) incorporates various modes of inhalation therapy. The response to treatments is dose dependent thus applying the most efficient device to administer the treatment is integral. Evaluation of the efficacy of nebulisation devices in the treatment of COPD is limited. Technological development in recent years has led to new devices that optimize lung deposition and reduce the time needed for treatment.

The aim of this study is to compare the vibrating mesh and jet nebuliser methods of delivering bronchodilator medication to patients hospitalised with an acute exacerbation of COPD, with respect to lung function and efficacy in spontaneously breathing patients.

Patients admitted to hospital with an exacerbation of COPD and prescribed regular nebulised bronchodilators (combined salbutamol 2.5mg and ipratropium 0.5mg) will be recruited to the study. On one occasion between day 3-7 of admission they will perform pulmonary function testing namely measurement of Forced Expiratory Volume in 1 second(FEV1), Forced Vital Capacity (FVC), Inspiratory Capacity (IC) and cough peak flow. They will also complete the Borg breathlessness score. Measurements will be recorded at baseline (pre-bronchodilator administration) and one hour post-nebulised bronchodilator.

Patients will be randomised to receive their nebulised bronchodilators via the standard hospital jet nebuliser or via a vibrating mesh nebuliser(Aerogen Solo).

Change in lung function and symptom measures between baseline and one-hour post nebulisation will be analysed to look for any significant difference between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Hospital Inpatients admitted with an acute exacerbation of COPD
* Age >40
* COPD Stage 2-4 moderate to severe (FEV1/FVC <0.70;FEV1<80%)
* History of physician-diagnosed COPD
* COPD exacerbation between day 2 and day 7 of admission

Exclusion Criteria:

* Confusion
* Significant hypoxia/unstable medical condition
* Allergy or contraindication to salbutamol and/or ipratropium
* Pneumonia
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory capacity (IC) | Baseline and One hour post nebulised bronchodilator

SECONDARY OUTCOMES:
Change in Forced expiratory volume in one second (FEV1) | Baseline and One hour post nebulised bronchodilator
Change in forced vital capacity (FVC) | Baseline and One hour post nebulised bronchodilator
Change in Borg breathlessness score | Baseline and One hour post nebulised bronchodilator
Change in Cough peak flow | Baseline and One hour post nebulised bronchodilator

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, Principal Investigator — RCSI
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No